CLINICAL TRIAL: NCT04848467
Title: COVID-19: A Phase 3, Randomized, Observer-blinded, Multicenter Clinical Study Evaluating the Immunogenicity, Safety, and Reactogenicity of the Investigational SARS-CoV-2 mRNA Vaccine CVnCoV, When Co-administered With a Licensed Quadrivalent Influenza Vaccine Versus Separate Administration of the Two Vaccines in Adults 60 Years of Age and Older
Brief Title: COVID-19: A Trial Studying the SARS-CoV-2 mRNA Vaccine CVnCoV to Learn About the Immune Response, the Safety, and the Degree of Typical Vaccination Reactions When CVnCoV is Given at the Same Time as a Flu Vaccine Compared to When the Vaccines Are Separately Given in Adults 60 Years of Age and Older
Acronym: CV-NCOV-011
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study cannot be conducted.
Sponsor: Bayer (Industry)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21819
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2 Infection; Coronavirus Disease 2019 (COVID-19)
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); COVID-19; mRNA Vaccine; SARS-CoV-2 mRNA Vaccine (CVnCoV); Quadrivalent influenza vaccine (QIV)
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Co-ad group (Experimental): Participants will receive CVnCoV at the same visit as QIV: first dose of CVnCoV and a dose of QIV in opposite arms at Day 1, the second dose of CVnCoV at Day 29, and a placebo injection at Day 57.
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine (CVnCoV); Biological: Quadrivalent influenza vaccine (QIV); Other: Placebo
- Group 2: Control group (Experimental): Participants will receive QIV and CVnCoV at two different visits: one dose of placebo and one dose of QIV in opposite arms at Day 1, the first dose of CVnCoV at Day 29 and the second dose of CVnCoV at Day 57.
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine (CVnCoV); Biological: Quadrivalent influenza vaccine (QIV); Other: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA Vaccine (CVnCoV) — Two intramuscular injections administered 28 days apart at a dose level of 12 μg mRNA.
  Other Names: CV07050101
Biological: Quadrivalent influenza vaccine (QIV) — One intramuscular injection as 0.5 mL. Each 0.5 mL dose will contain 15 μg haemagglutinin (HA) from each of the four influenza strains.
  Other Names: Influvac Tetra
Other: Placebo — One intramuscular injection as normal saline [0.9% NaCl].

SUMMARY:
The most recently discovered coronavirus (SARS-CoV-2) may cause illness in humans ranging from the common cold to serious illness, also referred to as Coronavirus disease 2019 (COVID-19). As of January 2021, there are only few authorized vaccines available for the prevention of COVID-19.

"CVnCoV" is a new SARS-CoV-2 messenger ribonucleic acid (mRNA) vaccine which is currently being developed for the prevention of COVID-19. The vaccine contains a molecule called mRNA which serves as an instruction manual for the cells in the body to produce a piece of protein from SARS-CoV-2 which activates the body´s defense system. The "CVnCoV" vaccine is injected into the muscle. After the injection, the body recognizes the protein as something that does not belong there. In this way the natural infection with the virus is imitated. The body activates immune cells to produce antibodies against the virus and creates specific immune cells called T cells.

"CVnCoV" is given in two doses separated by 28 days. In this study, the researchers will look at how well "CVnCoV" works when the first of the two doses is given together with a flu vaccine called seasonal quadrivalent influenza vaccine (QIV). They will also look at how well the flu vaccine works under these conditions. The QIV is injected into the muscle and is given as 1 dose. To see how well the participants' immune systems is activated by "CVnCoV" and QIV, the researches will measure the levels of specific antibodies against the viruses in the blood. Antibodies are proteins that allow the immune system to find and react to bacteria and viruses in the body. The researches will look into how safe the vaccination is and which type and degree of typical vaccination reactions are seen. To give "CVnCoV" and the flu vaccine together in the future when needed, e.g. during the flu season, would reduce the burden on the health system and on the patients.

Participants in this study are adults aged 60 years and older. In this study, participants are assigned to one of the two parallel groups of the same size. The assignment to either group is done by chance via a computer program. Participants in group 1 (Co-ad group) will receive CVnCoV at the same visit as QIV. Participants in group 2 (control group) will receive QIV and CVnCoV at two different visits. The Co-ad group will receive the first dose of CVnCoV and a dose of QIV in opposite arms at Day 1, the second dose of CVnCoV at Day 29, and a placebo injection, i.e. an injection that looks like a vaccination injection but does not contain vaccine, at Day 57. The control group will receive QIV and placebo in opposite arms at Day 1, the first dose of CVnCoV at day 29 and the second dose of CVnCoV at Day 57.

There will be five visits and four phone calls. During the study, the study team will take blood samples on four occasions to measure the antibodies against SARS-CoV-2, and nasopharyngeal swabs at 1 occasion. The physicians will do physical examinations at each visit. The participants will be asked how they are feeling and if they have any medical problems. They will, in addition, receive an electronic Diary to report medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participant of 60 years of age or older, at the time of signing the informed consent.
* Participants who are generally healthy. Note: healthy participant is defined as an individual who is in good general health, not having any symptomatic mental or physical disorder requiring regular or frequent medication. Subjects can be enrolled if the regular or frequent medication keeps the condition well controlled and asymptomatic with the treatment according to the investigator's discretion.
* Body mass index (BMI) within the range 18.0 and ≤35.0 kg m2 (inclusive).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Female participant of child-bearing potential.
* Use of any investigational or non-registered product (vaccine or drug) other than the study vaccine within 28 days or 5 times ½ life of the investigational product preceding the administration of the study vaccine, or planned use during the study period.
* Receipt of any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or planned receipt of any vaccine within 28 days of study vaccine administration.
* Receipt of any investigational, authorized or licensed, SARS-CoV-2 or other coronavirus vaccine prior to the administration of the CVnCoV study vaccine or planned receipt during the study.
* Receipt of an influenza vaccine within 6 months prior to enrollment in this study or planned receipt during the study.
* Receipt of any investigational or licensed lipid nanoparticles (LNP)-formulated mRNA vaccine prior to the administration of the study vaccine.
* Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to, corticosteroids, biologicals and methotrexate) for >14 days total within 6 months preceding the administration of study vaccine or planned use during the study. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 consecutive days or more. The use of inhaled, topical, intra-articular, intra-bursal corticosteroids is permitted.
* Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of the study vaccine.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including known human immunodeficiency virus infection, hepatitis B virus infection, or hepatitis C virus infection.
* Active cancer (under current treatment) or cancer requiring planned treatment in the past 5 years excluding non-melanoma skin cancer or cancers with excellent clinical prognosis (e.g. carcinoma in situ of the uterine cervix).
* History of known immune-deficiency disorders disease.
* History of angioedema (known C1 inhibitor deficiency).
* History of any anaphylactic reactions.
* Contraindications to administration of QIV as per current label, including history of severe allergic reactions (e.g., anaphylaxis) to any component of the QIV vaccine, including egg protein.
* Any known allergy to any component of CVnCoV or aminoglycoside antibiotics.
* History of confirmed SARS, MERS or COVID-19 disease or known exposure to an individual with confirmed COVID-19 disease or SARS-CoV-2 infection within 2 weeks prior to enrollment.
* Received or plan to receive 2021 inactivated seasonal influenza vaccine prior to or during the study and for the remaining of the 2021/2022 influenza season.
* Participants with a significant acute or chronic medical or psychiatric illness that, in the opinion of the investigator, precludes study participation (e.g., study participation may lay risks on the subject, renders the subject unable to meet the protocol requirements of the study, or may interfere with the reliability of the participant´s study readouts/results). These conditions may include severe and/or uncontrolled cardiovascular disease, gastrointestinal disease, liver disease, renal disease, respiratory disease, endocrine disorder, and neurological or psychiatric illnesses. However, those with well-controlled and those who are well-controlled and stable on their regular medication for their medical condition and have been so for the 12 weeks preceding the enrollment in this study can be included in the study.
* Participants with impaired coagulation or any bleeding disorder in whom an intramuscular injection or a blood draw is contraindicated.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Antibody titers for SARS-CoV-2 receptor binding domain (RBD) | 28 days after the second dose of CVnCoV
Hemagglutination inhibition (HI) titers for each of the 4 strains | 28 days after the QIV vaccination

SECONDARY OUTCOMES:
Number of participants seroconverting for SARS-CoV- 2 spike protein antibodies | 28 days after the second dose of CVnCoV
  Measured by enzyme-linked immunosorbent assay (ELISA).
SARS-CoV-2 spike protein-specific antibody levels in serum | 28 days after the second dose of CVnCoV
  Measured by enzyme-linked immunosorbent assay (ELISA).
Number of participants seroconverting for SARS-CoV- 2 neutralizing antibodies | 28 days after the second dose of CVnCoV
  Measured by an activity assay.
SARS-CoV-2 neutralizing antibody levels in serum | 28 days after the second dose of CVnCoV
Number of participants with seroprotection for serum antibodies against the 4 influenza vaccine strains | 28 days after the QIV dose
  Measured by hemagglutination inhibition (HI) assay.
Number of participants seroconverting for serum antibodies against the 4 influenza vaccine strains | 28 days after the QIV dose
  Measured by hemagglutination inhibition (HI) assay.
Serum antibody titers against the 4 influenza vaccine strains | 28 days after the QIV dose
  Measured by hemagglutination inhibition (HI) assay.
Number of participants with solicited local adverse events (AEs) of CVnCoV vaccine | Within 7 days after each study vaccination
Number of participants with solicited systemic AEs | Within 7 days after each study vaccination
Number of participants with unsolicited AEs | Within 28 days after each study vaccination
Number of participants with serious adverse event (SAEs) | Approximately 60 weeks
Number of participants with adverse event of special interest (AESIs) | Approximately 60 weeks

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.